CLINICAL TRIAL: NCT05131932
Title: Ablation of Esophageal Inlet Patches in Patients Referred for pH-Testing Due to Possible Extra-Esophageal Symptoms of Gastro-Esophageal Reflux Disease
Brief Title: Ablation of Esophageal Inlet Patches in Patients Referred for Bravo pH-Testing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0205-21-ASF
Record Dates: First submitted 2021-11-16; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: GERD; Cough; Metaplasia
MeSH Terms: conditions — Gastroesophageal Reflux; Cough; Metaplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inlet patch (Experimental): Patients found to have an inlet patch on upper endoscopy
  Interventions: Procedure: Endoscopic ablation of inlet patch
- Controls (No Intervention): Patients without an inlet patch on upper endoscopy

INTERVENTIONS:
Procedure: Endoscopic ablation of inlet patch — Endoscopic ablation of inlet patch using argon plasma coagulation (APC)
  Arms: Inlet patch

SUMMARY:
Patients with suspected extra-esophageal manifestations of gastro-esophageal reflux disease (GERD), such as cough, hoarseness, and globus, are often referred for pH testing. However, many of these symptoms may actually be due to an esophageal inlet patch. We aim to evaluate patients referred for pH testing to see if they have an inlet patch, to perform ablation of the inlet patch if detected, and then compare the outcomes of patients with an inlet patch who underwent ablation versus those without an inlet patch.

DETAILED DESCRIPTION:
Background The diagnosis of gastro-esophageal reflux disease (GERD) is difficult when patients present with extra-esophageal symptoms such as chronic cough, frequent throat clearing, globus sensation, sore throat, and hoarseness, as opposed to the traditional symptoms of heartburn and regurgitation.[1-4] These patients are often given a trial of proton pump inhibitors (PPIs) to see if their symptoms improve. They often undergo an upper endoscopy, which is usually unrevealing,[5] and they may be evaluated by other specialties such as otolaryngology and pulmonology. Eventually, some of these patients are referred for esophageal pH-testing to evaluate for objective evidence of acid reflux.

The symptoms of extra-esophageal GERD (EE-GERD) are not specific for GERD and many of them overlap with the symptoms from inlet patches, also known as heterotopic gastric mucosa.[6-7] Inlet patches consist of small areas of gastric mucosa in the upper esophagus that are capable of producing acid.[8-10] Studies in which inlet patches are endoscopically ablated have shown improvement in several extra-esophageal symptoms including globus sensation, sore throat, and cough.[11-15] As inlet patches are notoriously overlooked on upper endoscopy[16] and can cause many of the same symptoms as EE-GERD, we suspect that they may be responsible for the symptoms in some patients who are referred for pH-testing due to suspected EE-GERD. We believe that a careful inspection of the upper esophagus will reveal inlet patches that were missed on initial endoscopy and that ablation of these inlet patches will help improve the patients' symptoms more than the standard treatment for EE-GERD.

Aims The primary aim of this study is to evaluate the improvement in symptoms of patients referred for pH-testing for suspected EE-GERD that are treated with endoscopic ablation of an inlet patch versus those who receive standard PPI therapy. Secondarily, we seek to determine the prevalence of inlet patches in these patients with reportedly normal endoscopies, as well as percentage of patients in this group with a positive pH study.

Methods Patients referred for pH-testing due to symptoms of possible EE-GERD will be evaluated. These patients will have their prior medical history reviewed. Those with a prior normal endoscopy and inadequate response to PPI therapy will be included.

Patients' symptoms will be assessed via a questionnaire across 8 domains including 6 symptoms of possible EE-GERD and 2 subjective scores of how the symptoms are affecting their lives (see Questionnaire below). A visual Likert scale from 0 to 10 will be used. An overall symptom score will be calculated based on the results of the 8 individual domains.

Patients will then undergo an upper endoscopy. During the endoscopy, care will be taken to assess for possible inlet patches. Advanced imaging techniques such as i-scan imaging will be used to aid in the detection of inlet patches. If one or more inlet patches are found, the number, size, and shape will be recorded, and it will be biopsied for histological confirmation. The inlet patch will then be ablated via the use of argon plasma coagulation (APC) as has been performed in prior studies.[11-13] During the endoscopy, a Bravo pH capsule will also be placed per standard protocol to complete a 48-hour pH study. The Bravo data will be interpreted according to standard procedure with a positive study defined as an elevated DeMeester score on either study day. All studies will be performed off of anti-acid medications such as PPIs.

The patients' symptoms will be re-assessed at 2 and 6 months following the endoscopy. This will be performed via telephone interviews with the patients completing the same symptom assessments as prior to the endoscopy. Changes in their medications and treatment as a result of the Bravo pH study results will also be evaluated.

The primary end point will be the symptom improvement in overall score in patients who underwent ablation of inlet patches versus those without inlet patches.

Inclusion Criteria

* Adult patients (age 18 and above)
* Referred for pH-testing for evaluation of possible EE-GERD
* Prior upper endoscopy performed
* Prior trial of PPI with an inadequate response Exclusion Criteria
* Patients who do not give consent
* Patients with abnormalities on their prior endoscopy including a significant hiatal hernia (>3 cm) or significant erosive esophagitis (Los Angeles class B or greater)
* Patients who did not fail a prior trial of PPI therapy Anticipated number of subjects: 100

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 and above)
* Referred for pH-testing for evaluation of possible extraesophageal-GERD
* Prior upper endoscopy performed
* Prior trial of PPI with an inadequate response

Exclusion Criteria:

* Patients who do not give consent
* Patients with abnormalities on their prior endoscopy including a significant hiatal hernia (>3 cm) or significant erosive esophagitis (Los Angeles class B or greater)
* Patients who did not fail a prior trial of PPI therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Symptoms 6 months after procedure | 6 months after procedure
  The overall symptoms score

SECONDARY OUTCOMES:
Symptoms 2 months after procedure | 2 months after procedure
  The overall symptoms score

IPD SHARING:
Plan to Share IPD: No
IPD will be kept securely at the medical center

REFERENCES:
- [Background] Vaezi MF, Katzka D, Zerbib F. Extraesophageal Symptoms and Diseases Attributed to GERD: Where is the Pendulum Swinging Now? Clin Gastroenterol Hepatol. 2018 Jul;16(7):1018-1029. doi: 10.1016/j.cgh.2018.02.001. Epub 2018 Feb 7. PMID 29427733
- [Background] Madanick RD. Extraesophageal presentations of GERD: where is the science? Gastroenterol Clin North Am. 2014 Mar;43(1):105-20. doi: 10.1016/j.gtc.2013.11.007. Epub 2013 Dec 28. PMID 24503362
- [Background] Ghisa M, Della Coletta M, Barbuscio I, Marabotto E, Barberio B, Frazzoni M, De Bortoli N, Zentilin P, Tolone S, Ottonello A, Lorenzon G, Savarino V, Savarino E. Updates in the field of non-esophageal gastroesophageal reflux disorder. Expert Rev Gastroenterol Hepatol. 2019 Sep;13(9):827-838. doi: 10.1080/17474124.2019.1645593. Epub 2019 Jul 22. PMID 31322443
- [Background] Sidhwa F, Moore A, Alligood E, Fisichella PM. Diagnosis and Treatment of the Extraesophageal Manifestations of Gastroesophageal Reflux Disease. Ann Surg. 2017 Jan;265(1):63-67. doi: 10.1097/SLA.0000000000001907. PMID 27455157
- [Background] Zullo A, Fiorini G, Bassotti G, Bachetti F, Monica F, Macor D, Paoluzi OA, Scaccianoce G, Portincasa P, De Francesco V, Lorenzetti R, Saracino IM, Pavoni M, Vaira D. Upper Endoscopy in Patients with Extra-Oesophageal Reflux Symptoms: A Multicentre Study. GE Port J Gastroenterol. 2020 Aug;27(5):312-317. doi: 10.1159/000505581. Epub 2020 Feb 4. PMID 32999903
- [Background] von Rahden BH, Stein HJ, Becker K, Liebermann-Meffert D, Siewert JR. Heterotopic gastric mucosa of the esophagus: literature-review and proposal of a clinicopathologic classification. Am J Gastroenterol. 2004 Mar;99(3):543-51. doi: 10.1111/j.1572-0241.2004.04082.x. PMID 15056100
- [Background] Ciocalteu A, Popa P, Ionescu M, Gheonea DI. Issues and controversies in esophageal inlet patch. World J Gastroenterol. 2019 Aug 14;25(30):4061-4073. doi: 10.3748/wjg.v25.i30.4061. PMID 31435164
- [Background] Galan AR, Katzka DA, Castell DO. Acid secretion from an esophageal inlet patch demonstrated by ambulatory pH monitoring. Gastroenterology. 1998 Dec;115(6):1574-6. doi: 10.1016/s0016-5085(98)70038-1. PMID 9834287
- [Background] Hamilton JW, Thune RG, Morrissey JF. Symptomatic ectopic gastric epithelium of the cervical esophagus. Demonstration of acid production with Congo red. Dig Dis Sci. 1986 Apr;31(4):337-42. doi: 10.1007/BF01311666. PMID 3956328
- [Background] Nakajima H, Munakata A, Sasaki Y, Yoshida Y. pH profile of esophagus in patients with inlet patch of heterotopic gastric mucosa after tetragastrin stimulation. An endoscopic approach. Dig Dis Sci. 1993 Oct;38(10):1915-9. doi: 10.1007/BF01296118. PMID 8404414
- [Background] Meining A, Bajbouj M, Preeg M, Reichenberger J, Kassem AM, Huber W, Brockmeyer SJ, Hannig C, Hofler H, Prinz C, Schmid RM. Argon plasma ablation of gastric inlet patches in the cervical esophagus may alleviate globus sensation: a pilot trial. Endoscopy. 2006 Jun;38(6):566-70. doi: 10.1055/s-2006-925362. PMID 16802267
- [Background] Bajbouj M, Becker V, Eckel F, Miehlke S, Pech O, Prinz C, Schmid RM, Meining A. Argon plasma coagulation of cervical heterotopic gastric mucosa as an alternative treatment for globus sensations. Gastroenterology. 2009 Aug;137(2):440-4. doi: 10.1053/j.gastro.2009.04.053. Epub 2009 May 4. PMID 19410576
- [Background] Klare P, Meining A, von Delius S, Wolf P, Konukiewitz B, Schmid RM, Bajbouj M. Argon plasma coagulation of gastric inlet patches for the treatment of globus sensation: it is an effective therapy in the long term. Digestion. 2013;88(3):165-71. doi: 10.1159/000355274. Epub 2013 Oct 18. PMID 24157960
- [Background] Dunn JM, Sui G, Anggiansah A, Wong T. Radiofrequency ablation of symptomatic cervical inlet patch using a through-the-scope device: a pilot study. Gastrointest Endosc. 2016 Dec;84(6):1022-1026.e2. doi: 10.1016/j.gie.2016.06.037. Epub 2016 Jul 1. PMID 27373671
- [Background] Kristo I, Rieder E, Paireder M, Schwameis K, Jomrich G, Dolak W, Parzefall T, Riegler M, Asari R, Schoppmann SF. Radiofrequency ablation in patients with large cervical heterotopic gastric mucosa and globus sensation: Closing the treatment gap. Dig Endosc. 2018 Mar;30(2):212-218. doi: 10.1111/den.12959. Epub 2017 Oct 3. PMID 28884487
- [Background] Peitz U, Vieth M, Evert M, Arand J, Roessner A, Malfertheiner P. The prevalence of gastric heterotopia of the proximal esophagus is underestimated, but preneoplasia is rare - correlation with Barrett's esophagus. BMC Gastroenterol. 2017 Jul 12;17(1):87. doi: 10.1186/s12876-017-0644-3. PMID 28701149